CLINICAL TRIAL: NCT03775239
Title: Mindfulness as Treatment of Sexological Problems: A Randomized, Controlled Pilot Study of Mindfulness in Sex Therapy and Intimate Relationships (MSIR) in the Treatment of Sexual Dysfunctions
Brief Title: Mindfulness as Treatment of Sexological Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Den Owesenske Fond (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-18017600
Record Dates: First submitted 2018-09-14; First posted 2018-12-13 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-12

CONDITIONS: Sexual Dysfunction; Sexual Dysfunctions, Psychological; Sexual Dysfunctions, Physiological
Keywords: Desire dysfunction; Erectile dysfunction; Orgasm dysfunction; Sexual pain; Hyper sexuality; Mindfulness
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Erectile Dysfunction | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-as-usual (Other): Those who are randomly selected to treatment-as-usual will receive a minimum of 6 sessions at Sexological Clinic.
  Interventions: Behavioral: Treatment-as-usual
- Treatment-as-usual + MSIR (Other): Those who are randomly selected to receive Mindfulness in Sex Therapy and Intimate Relationships (MSIR) will first receive 6 weeks of mindfulness followed by treatment-as-usual. The intervention will take place at Sexological Clinic.
  Interventions: Behavioral: Mindfulness in Sex Therapy and Intimate Relationships (MSIR); Behavioral: Treatment-as-usual

INTERVENTIONS:
Behavioral: Mindfulness in Sex Therapy and Intimate Relationships (MSIR) — Mindfulness is a mental discipline inviting intentional, non-judgmental attending of the stream of experience. Mindfulness can be seen as an adjunct to sexual therapy. Firstly, it is a way of teaching the patients and the couples to carry out sensate focus so that it can achieve its goals. Beyond this, Mindfulness may invite a stance to one's own and a partner's physical and emotional experience that is more widely beneficial. The MSIR intervention was originally developed from the Mindfulness Based Cognitive Therapy (MBCT) protocol and consists of:
  Week 1: Moving into the Body Week 2: Sensing & Exploring Week 3: Avoidance & Intimacy- Midway individual session. Week 4: Recognising our automatic mind Week 5: Spacious Awareness Week 6: Expanding new learning
  Arms: Treatment-as-usual + MSIR
Behavioral: Treatment-as-usual — The current treatment in Sexological Clinic is an eclectic, synthetic therapy form conducted by psychiatrists, other medical doctors, psychologists and bodytherapists.
  In order to implement the bio-psycho-social character of sexual dysfunctions, the current treatment takes advantage of different elements from different therapy forms combined with pharmacological treatment if necessary.
  The integrated treatment combines elements from therapy's such as cognitive behavioural therapy (CBT), psychodynamic therapy and systemic therapy together with Master and Johnson's sensate focus training, body exercises training as pelvis floor exercises, introduction of sexual aids and if necessary pharmacological treatment. The therapy can be individual treatment, couple therapy (marital therapy) or group therapy.

SUMMARY:
The primary aim of this study is to test Mindfulness in Sex Therapy and Intimate Relationships (MSIR) as an add-on treatment to sex therapy in a clinical sample of patients referred with sexual problems, controlling for time effect, with a treatment as usual activity group.

The secondary aim is to investigate the effect of MSIR alone on sexual dysfunction compared to treatment-as-usual (TAU).

It is hypothesized that the MSIR group, in preceding the usual TAU intervention, will achieve greater benefits in relation to sexual functioning outcomes as measured by subjective and objective measures. The investigators expect that MSIR will help the patients to cultivate accept and body awareness, which will create a wider sense of safety and stability that might help integrating the assistant provided by the traditional approach to the treatment of sexual dysfunctions. It is hypothesized that the intervention (MSIR+TAU) reduces the amount of TAU sessions needed in order to achieve a benefit in terms of the patient's sexual dysfunction.

It is furthermore, hypothesized that the intervention (MSIR) alone will have a positive effect on the sexual dysfunction.

The research project outlines a pragmatic pilot randomized control trial to evaluate MSIR treatment as an add-on to the treatment-as-usual (TAU) compared to TAU for sexual difficulties in men and women.

DETAILED DESCRIPTION:
BACKGROUND:

Prevalence of sexual dysfunction is high, although estimates are variable. For men, the reported level of sexual difficulty, taking all conditions into account, is around 33% or up to 46%. For women, the reported level of sexual difficulty is higher, with estimates up to around 66%. Sexual dysfunctions are associated with a negative impact on the quality of life in both men and women and there is therefore a need for effective treatments.

AIM:

The primary aim of this study is to test Mindfulness in Sex Therapy and Intimate Relationships (MSIR) as an add-on treatment to sex therapy in a clinical sample of patients referred with sexual problems, controlling for time effect, with a treatment as usual activity group.

The secondary aim is to investigate the effect of MSIR alone on sexual dysfunction compared to treatment-as-usual (TAU).

It is hypothesized that the MSIR group, in preceding the usual TAU intervention, will achieve greater benefits in relation to sexual functioning outcomes as measured by subjective and objective measures. The investigators expect that MSIR will help the patients to cultivate accept and body awareness, which will create a wider sense of safety and stability that might help integrating the assistant provided by the traditional approach to the treatment of sexual dysfunctions. It is hypothesized that the intervention (MSIR+TAU) reduces the amount of TAU sessions needed in order to achieve a benefit in terms of the patient's sexual dysfunction.

It is furthermore, hypothesized that the intervention (MSIR) alone will have a positive effect on the sexual dysfunction

METHODS:

The present study will take form as a feasibility study and is seen as a pilot study which will provide a view on MSIR's effectiveness in the natural environment of Sexological Clinic, Psychiatric Centre Copenhagen.

The research project outlines a pragmatic randomized control trial to evaluate MSIR treatment as an add-on to the treatment-as-usual (TAU) compared to TAU for male and female sexual difficulties. The participants will be drawn from Sexological Clinic's patients referred with sexual problems as decreased desire, erectile dysfunction, orgasmic/ejaculatory dysfunction or hypersexuality.

30 patients will be included; 15 in the MSIR group and 15 as controls. The investigators aim for an equal number of men and women in each group. To follow the methodology of a pragmatic design, the inclusion and exclusion criteria will be kept at a minimum.

MEASURES:

Validated questionnaires will measure the main dependent variables: sexual functioning (FSFI, FSDS, IIEF), mindfulness (TMS, MAIA, FFMQ) and number of sessions of treatment completed. Descriptive variables are SCL-10, well-being (WHO-5) and sociodemographic questionnaire. The questionnaires will be handed out before the beginning of the treatment, after 3 sessions, after 6 sessions, after 9 sessions, in the end of the treatment and then after 6 months of follow-up.

STATISTICS:

Baseline characteristics of the two groups will be compared as appropriate, using independent samples t-test for continuous variables, Kruskal-Wallis and chi-square for categorical variables. The second step is calculating the effect size for change in each dimension for each group using Cohens' d. The statistically significant level p < 0.05 (two sides) will be used.

ETHICAL CONSIDERATIONS:

The trial is approved by the Regional Ethics Committee in the Capital Region of Denmark and the Danish Data Protection agency.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 20-65 years referred to Sexological Clinic and diagnosed with sexual dysfunction (desire dysfunction, erectile dysfunction, orgasm dysfunction, sexual pain or hyper sexuality).

* After assessment, being allocated to individual or couple therapy for their sexual dysfunction. The partner will be included in case of couples therapy
* Allocated to a minimum of 6 treatment sessions in TAU after assessment
* Giving informed consent
* Being able to read, write, speak and understand the Danish language.

Exclusion Criteria:

* Assessed for group therapy
* Cannot participate at the scheduled MSIR session due for practical reasons
* Having experienced sexual trauma in the past, suffering from mental illness, severe somatic disease and/or addiction
* Withdrawing their informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
The Sexual Function Questionnaire for Females & Males (CSFQ-14-F/M) | Change from baseline CSFQ score to 6 month follow-up CSFQ score
  The CSFQ is a 14 item self-report inventory which measures sexual functioning on a 5 point likert scale. The questionnaire comprises: a 5 scale structure consistent with the original (longer) CSFQ - Desire/Frequency, Desire/Interest, Arousal/Excitement, Orgasm/Completion, Pleasure, The questionnaire has a high degree of internal consistency as a whole (Cronbach's alpha = 0.90 for females and 0.89 for males) and for the individual scales (all were between 0.68 and 0.84, except the male orgasm/completion scale, 0.59). Good scale coherency and discrimination was demonstrated by highly significant mean difference scores between the CSFQ and control groups.
Female Sexual Function Index (FSFI) | Change from baseline FSFI score to 6 month follow-up FSFI score
  The Female Sexual Function Index (FSFI) is a validated 19-item multidimensional self-report instrument for the assessment of female sexual function that comprise a full scale and six subscales (desire, arousal, lubrication, orgasm, satisfaction and pain). It measures the overall sexual function through either 0-5 or 1-5-point Likert scales. A higher score represents better sexual function. A score equal to or below 26.55 points represents a risk of sexual dysfunction. The FSFI has shown test-retest reliability (r=0,75-0,86). The scale is recommended for clinical practice as a measure of symptoms severity in women who have been sexually active in the prior 4 weeks51 and is the golden standard when measuring sexual function in women
Female Sexual Distress Scale (FSDS) | Change from baseline FSDS score to 6 month follow-up FSDS score
  The Female Sexual Distress Scale (FSDS) is a validated 12-item self-administered questionnaire, developed to measure sexually related personal distress in women. Lower scores represent less sexual distress. Scores equal to or above 15 points indicates sexually related distress.
The International Index of Erectile Function (IIEF) | Change from baseline IIEF score to 6 month follow-up IIEF score
  The IIEF is a validated self-administered 15-item questionnaire that asses male sexual function. The IIEF-questionnaire seeks to detect treatment-related changes in patients with erectile functions and is the golden standard. The IIEF comprises a full scale and five subdomains (erectile function, orgasmic function, sexual desire, intercourse satisfaction and overall satisfaction). A low score represents worse sexual function. The questionnaire comprises a full scale and five subdomains. The subdomains are; erectile function; orgasmic function; sexual desire; intercourse satisfaction; and overall satisfaction).
Bothered by Problem (VAS) | Change from baseline VAS score to 6 month follow-up VAS score
  Single-item distress scale measuring on a Likert scale from 1-10 (10 is most distressed) distress by the problem which the person sought help for. "How bothered are you at this time of the problem you are/were seeking for help for?"

SECONDARY OUTCOMES:
The Five Facet Mindfulness Questionnaire (FFMQ) | 1 time a week after mindfulness session up to 8 weeks
  The FFMQ is a 39-item selfreport scale that measures levels of dispositional mindfulness in everyday life across the five facets: observing, describing, acting with awareness, non-judging and non-reactivity.
The Multidimensional Assessment of Interoceptive Awareness (MAIA) | Week 0, week 3,6,9,month 6
  The MAIA is a self-report public domain questionnaire developed. It is a 32-item multidimensional instrument that assesses eight concepts. The scale has been confirmed as a valuable source in understanding clinical outcomes, as the MAIA is concerned with understanding a large scope of medical and psychological conditions.
World Health Organization 5 Wellbeing Questionnaire (WHO-5) | Week 0, week 3,6,9,month 6
  The WHO-5 is a self-administered 5 item questionnaire assessing the degree of positive well-being during the past 2 weeks on a six-point Likert scale graded from 0 (at no time) to 5 (all of the time), and the total score ranges from 0 to 25, with high scores indicating an increased sense of well-being. It has been shown to have good internal reliability (Cronbach's Alpha = 0.89), external concurrent validity and discriminatory validity as a screening tool for depression (p<0.001) in older people, diabetic patients and a general outpatient sample.
The Symptom Checklist (SCL-10) | Week 0, week 3,6,9,month 6
  The SCL-10 is a brief version developed from the SCL-90 questionnaire that measures mental or affective distress. The SCL-10 is well validated to measure psychological distress. The SCL-10 has been translated into Danish and is routinely used when measuring the effect of psychotherapeutic intervention. The questionnaire uses a 5-point Likert scale rate ranging from 0 (not at all) to 4 (extremely) and measures the past two weeks.

OTHER OUTCOMES:
Questionnaire to collect individual demographic data | Week 0 and month 6.
  The demographic questionnaire will entail questions concerning date of birth, gender, relationship status, medication, education and occupation. These demographic questions can through statistical analysis help us identify a potential pattern of who is more susceptible for treatment and if there are any correlations.

CONTACTS AND LOCATIONS:
Locations (1):
- Sexological Clinic, Copenhagen, Denmark